CLINICAL TRIAL: NCT04678336
Title: Phase 1 Study of Lentivirally Transduced T Cells Engineered to Contain Anti-CD123 Linked to TCRζ and 4-1BB Signaling Domains in Pediatric Subjects With Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: CD123 Redirected T Cells for AML in Pediatric Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 834675 (19CT011)
Record Dates: First submitted 2020-10-22; First posted 2020-12-21 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia, Pediatric; Acute Myeloid Leukemia, Refractory
Keywords: refractory; relapsed; Acute; Myeloid; leukemia; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Leukemia | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): CART123 cells; cyclophosphamide; fludarabine
  Interventions: Biological: CART123 cells; cyclophosphamide; fludarabine

INTERVENTIONS:
Biological: CART123 cells; cyclophosphamide; fludarabine — CART123 cells following lymphodepleting chemotherapy in pediatric patients with relapsed/refractory AML. Subjects will be treated with a single IV dose of CART123 cells on Day 0.
  Other Names: T Cells Containing Anti-CD123 Signaling Domains

SUMMARY:
Phase 1 open-label study to evaluate the safety of intravenously administered, lentivirally transduced T cells expressing anti-CD123 chimeric antigen receptors expressing tandem TCRζ and 4-1BB (TCRζ /4-1BB) costimulatory domains in pediatric subjects with relapsed/refractory Acute Myeloid Leukemia (AML).

DETAILED DESCRIPTION:
This is a Phase 1 study designed to evaluate the safety, feasibility, and preliminary efficacy of CART123 cells in pediatric subjects with relapsed/refractory Acute Myeloid Leukemia (AML). The study was originally designed to evaluate these primary endpoints at a single CART123 dose level (2x106 CART123 cells/kg). This dose level was selected based on experience in an adult trial using this investigational product in relapsed/refractory AML patients (NCT03766126).

As of Protocol Amendment V6, the study design has been converted into a 3+3 dose escalation design in order to further explore the safety of CART123 cells in the target disease population, and determine a maximum tolerated dose (MTD). The initial dose level (2x106 CART123 cells/kg) will be retrospectively identified as Dose Level 1 (DL1), and up to two new dose levels of CART123 cells will now be evaluated as follows:

* Dose Level 1 (DL1): 2x106 CART123 cells/kg

  o <DL1 Fully Enrolled as of Protocol Amendment V6>
* Dose Level 2 (DL2): 5x106 CART123 cells/kg
* Dose Level 3 (DL3): 1x107 CART123 cells/kg

Dose Level 1 (DL1) was fully evaluated as of Protocol Amendment V6. Dose Level 2 (DL2) and Dose Level 3 (DL3) will be evaluated as follows:

* Dose Level 2 (N = 3-6):

  * If 1 DLT/3 subjects occurs, 3 additional DLT-evaluable subjects will enrolled at this dose level.
  * If 0 DLT/3 subjects or 1 DLT/6 subjects occur, DL2 safety data will be submitted to the DSMB for review. DSMB approval must be received in order to advance to Dose Level 3 (DL3).
  * If 2 DLTs occur at any time, additional enrollment on this study will be paused to allow for further investigation.
* Dose Level 3 (N = 3-6):

  * If 1 DLT/3 subjects occurs, 3 additional DLT-evaluable subjects will be enrolled at this dose level.
  * If 0 DLT/3 subjects, 3 additional DLT-evaluable subjects will be enrolled at this dose level to further evaluate safety and allow for MTD determination.
  * If 2 DLTs occur at any time, enrollment at this dose level will be stopped. If fewer than 6 evaluable subjects were infused at DL2, additional subjects will be enrolled at that dose level to reach a minimum of 6 DLT-evaluable subjects for MTD determination.

The DLT observation period is 28 days post-CART123 cell infusion (Day 0). In order to allow for appropriate monitoring/assessment of toxicities, study treatment in the 1st and 2nd subjects at each dose level must be staggered by at least 28 days, such that the next subject will not receive treatment (lymphodepleting chemotherapy plus CART123 cells) until the previous subject has completed their Day 28 safety follow-up visit. If there are no emergent safety concerns identified in the first subject infused, study treatment for subsequent subjects at that same dose level do not need to be staggered and may occur sequentially without additional staggering requirements. Formal DLT evaluations will be performed after the 3rd evaluable subject at each dose level reaches the Day 28 safety follow-up visit. These formal DLT evaluations will allow for a formal decision regarding dose level progression, expansion, or dose de-escalation. Formal DLT evaluations will be determined by the Clinical PI and Sponsor Medical Director in accordance with the definition in the protocol. The MTD is defined as the highest dose at which 0 or 1 DLT occurs in 6 evaluable subjects.

It is recommended that subjects with marrow aplasia at Day 28+/-5 undergo an allogeneic hematopoietic cell transplantation (alloHCT) as a rescue strategy. If required, this procedure will be performed as part of routine care, outside of the scope of this research study; however, subjects will continue to be followed onstudy. All subjects must, therefore, have a previously identified stem cell donor as part of their eligibility to participate in this study. All subjects will be followed monthly for up to 6 months after the CART123 cell infusion (Day 0). Thereafter, subjects will be transitioned into LTFU for up to 15 years post infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥ 1 and ≤ 29 years of age at time of consent.
2. AML in second or greater relapse, post-transplant relapse, or chemotherapy-refractory disease. Specifically:

   1. Second or greater relapse defined as flow cytometric confirmation of myeloid leukemia of at least 0.1% after second documented complete remission; OR
   2. Any detectable disease post-allogeneic transplant with flow cytometric confirmation (MRD) of myeloid leukemia of at least 0.1% (as confirmed by Hematologics); OR
   3. Refractory disease, defined as persistent bone marrow involvement with >5% blasts after two courses of induction chemotherapy for patients at initial presentation or >5% bone marrow blasts after one course of re-induction chemotherapy for patients who have relapsed after previously achieving a CR.
3. Subjects must have a suitable stem cell donor identified with projected ability to proceed to transplant within 6-8 weeks of CART123 infusion.
4. Adequate organ function defined as:

   1. A serum creatinine based on age/gender
   2. Adequate liver function

   i. ALT ≤ 5 x ULN

   ii. Total bilirubin ≤ 3 x ULN

   iii. ALT and/or bilirubin results that exceed this range are acceptable if, in the opinion of the physician-investigator (or as confirmed by liver biopsy), the abnormalities are directly related to AML infiltration of the liver.

   c. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and < Grade 3 hypoxia; DLCO ≥ 40% (corrected for anemia) if PFTs are clinically appropriate as determined by the treating investigator

   d. Left Ventricular Shortening Fraction (LVSF) ≥ 28% or Ejection Fraction (LVEF) ≥ 45% confirmed by ECHO, or adequate ventricular function documented by a scan or a cardiologist. In cases where quantitative assessment of LVSF/LVEF is not possible, a statement by the cardiologist that the ECHO shows qualitatively normal ventricular function will suffice.
5. Adequate performance status defined as Lansky or Karnofsky score ≥ 50
6. Signed informed consent must be obtained.
7. No contraindications for leukapheresis (unless apheresis product previously acquired).
8. Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion Criteria:

1. Pregnant or lactating (nursing) women.
2. Patients with relapsed AML with t(15:17).
3. Patients < 6 months from alloHSCT.
4. HIV infection.
5. Active hepatitis B or hepatitis C infection.
6. Active acute or chronic graft-versus-host disease (GVHD) requiring systemic therapy
7. Patients requiring chronic treatment with systemic steroids or immunosuppressant medications. Low-dose physiologic replacement therapy with corticosteroids, topical steroids and inhaled steroids are acceptable. For additional details regarding use of steroids and immunosuppressant medications (including washout requirements prior to CAR T cell administration).
8. Any uncontrolled active medical disorder that would preclude participation as outlined.
9. Uncontrolled active infection
10. Subjects with CNS3 disease that is progressive on therapy or with CNS parenchymal lesions that may increase the risk of CNS toxicity. Subjects with adequately treated CNS leukemia are eligible.
11. Known history of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).
12. Patients with any prior history of myeloproliferative neoplasm.
13. Patients with somatic JAK2 V617F mutation by PCR or next generation sequencing.

Ages: 1 Year to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of CART123 in AML subjects | 5 Years
  * Occurrence of adverse events that are possibly, probably, or definitely related to CART123 cells
  * Occurrence of dose-limiting toxicities (DLTs) and determination of Maximum Tolerated Dose (MTD)

SECONDARY OUTCOMES:
Evaluate study feasibility | 15 Years
  • Proportion of enrolled subjects that screen fail; Proportion of enrolled subjects who receive study treatment.
Evaluate manufacturing feasibility | 15 Years
  • Frequency of product release failures; Occurrence of dose failures (inability to meet targeted dose).
Describe preliminary efficacy | 15 Years
  * Reduction of blast count in the peripheral blood and marrow using standard clinical criteria (CBC with differential count, marrow aspirate with differential count) and flow cytometry
  * Overall Response Rate (ORR) at 28 +/- 5 days
  * Overall survival (OS)
  * Progression-free survival (PFS)
  * Duration of Response (DOR)
Evaluate the need for rescue alloHCT | 15 Years
  • Percentage of subjects proceeding to alloHCT (or second allogeneic HCT)

OTHER OUTCOMES:
Determine persistence and trafficking of CART123 cells | 15 Years
  * The duration of in vivo survival of CART123 cells ("persistence") is defined as the period of time above the limit of detection of Q-PCR for peripheral blood CART123 transgene sequences and/or flow cytometry for scFv surface expression.
  * Trafficking will be determined by performing Q-PCR and flow cytometry as above on bone marrow samples and/or other tissue biopsies as clinically indicated
Analyze CART123 bioactivity | 15 Years
  • Multiplex cytokine analysis will be performed at multiple time points; if CRS develops, cytokine analysis will be performed from samples collected during CRS until its clinical resolution to follow the kinetics of cytokines longitudinally. This analysis will be batched and not available in real time or for clinical decisions.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No